CLINICAL TRIAL: NCT04763382
Title: The Effect of Nursing Interventions for Clean Intermittent Catheterization on Knowledge / Skills, Coping / Adaptation, Anxiety and Infection Development in Child Caregivers
Brief Title: The Effect of Nursing Interventions for Clean Intermittent Catheterization Caregivers and Child
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Canan Sari, Principal Investigator, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nurse_clean intermittent cat.
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Intermittent Urethral Catheterization; Spinal Dysraphism; Urinary Tract Infections
Keywords: Anxiety; Child; Nurses; Urinary Tract Infection; Intermittent Urethral Catheterization; Quality of Life; Caregivers; Mobile Applications; Smartphone
MeSH Terms: conditions — Spinal Dysraphism; Urinary Tract Infections; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The caregivers in experimental group of study were given health training on CIC application, and after the training, the guide booklet was delivered to the participants, the android phone application. After discharge of three urinalysis, three phone calls and home visit. The data collection tools applied to aregivers in experimental group as a pre-test were also applied post-test and retention test. The same data collection tools were applied to control group for pre-test. The caregivers in the control group were not trained, android applications were not installed on their phones, home visits. With the routine practice given in the hospital, he was provided with CIC training. However, one month after discharge, he was asked to give urinalysis once a month for three consecutive months. Urinalysis was taken three times in total. Data collection tools, which were applied as a pre-test when they gave the second urinalysis, were applied again as a post-test.
Masking Description: Because the initiative of the study is based on education. While obtaining informed consent, the purpose and content of the study were explained to the participants. For this reason, the trainees know that they are in the experimental group, and those who do not receive training in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental grups: Training of caregivers (Other): 1. Application of data collection:
     Tools as pre-test, post-test and retention test to participants in the experimental group,
  2. Education:It includes the training given to the caregivers in the experimental group, delivery of the guide booklet at the end of the training
  3. Android phone application: Installing on the phones of the caregivers in the experimental group of the android application, which includes the frequency of CIC application, the CIC application process steps and hospital appointments, created by the nurse for the caregivers in the experimental group and the software is made by the computer engineer.
  4. One home visit and three phone calls were made in order to solve the problems that the caregivers in the experimental group experienced with the use of CIC or android use.
  5. Urinalysis for children who are inserted and put into the study:All participants in the study were asked to give urine tests three times with an interval of one month after discharge.
  Interventions: Other: experimental group: Training of caregivers
- Control: Control grups (Other): 1. As in the experimental group, the caregivers in the control group were pre-tested and post-tested using data collection tools.
  2. No intervention was made to the caregivers in the control group.
  3. However, caregivers in the control group performed urinalysis three times with an interval of one month after discharge.
  Interventions: Other: Control gruop

INTERVENTIONS:
Other: experimental group: Training of caregivers — Pre-test, post-test, retention test, education, guide booklet delivery, android application installation and urinalysis
  Arms: Experimental grups: Training of caregivers
Other: Control gruop — Pre-test, post-test and urinalysis
  Arms: Control: Control grups

SUMMARY:
In neurogenic or non-neurogenic bladder disorders, the removal process after the catheter is inserted into the bladder and the urine has been drained is called Clean intermittent catheterization (CIC). After 1972, Lapides started using CIC in the treatment of people who cannot empty their bladder on their own. The decision to apply CIC to patients is made by the doctor. After CIC application, patients's increase body image, self-confidence development and quality of life. CIC application to children is done by caregivers. CIC use has negative effects as well as positive effects for patients. If the caregiver has not received enough training about CIC application and does not pay attention to CIC performing hours and procedure steps, urinary tract infection can be seen in children. Common urinary tract infections in children cause permanent kidney damage. Studies conducted to prevent complications that may develop in patients using CIC emphasize the importance of patient education. The aim of this study is to evaluate the effect of based on the roy adaptation theory supported android phone application CIC training, on the knowledge / skills, coping / adaptation and anxiety level of caregivers and the development of urinary tract infection in children.

DETAILED DESCRIPTION:
Background: It is the bladder, one of the organs with important functions in the urinary system. However, the bladder sometimes cannot work effectively as a result of neurological and sometimes non-neurological reasons. After this situation, urine in the bladder should be emptied. The bladder is one of the most frequently used organs in the urinary system. In neurogenic or non-neurogenic bladder disorders, the process of entering the bladder with a catheter in clean conditions, evacuating urine, and then removing the catheter is called Clean Intermittent Catheterization (CIC). CIC has been used by patients for nearly 40 years. CIC is one of the effective methods used to protect the urinary system, especially in children with Spina Bifida and people with urinary system problems. CIC application to children is done by caregivers. In the education of caregivers who have to apply CIC to their child the role of nurse to become more and more important. The aim of this study is to evaluate the effect of based on the roy adaptation theory supported android phone application CIC training, on the knowledge / skills, coping / adaptation and anxiety level of caregivers and the development of urinary tract infection in children.

Metod: The universe of the study consisted of the patients and their caregivers who were decided to perform CIC by Karadeniz Technical University Farabi Hospital Pediatric Nephrology Department. In order to determine the sample of the study, the test power in power analysis was calculated with the G * Power 3.1 program. 95% confidence interval in determining the strength of the study; With 5% significance level and 0.50 effect size a total of 36 patients (df = 1; F = 4.130). 36 conforming patients were divided into experimental and control groups for a single- blind randomized control. The data will be collected using the introductory information form, the CIC application knowledge and skills form, based on North American Association of Nursing Diagnoses (NANDA) nursing diagnoses and Psychosocial Adaptation Area of Roy Adaptation Model form, Coping and Adaptation Scale and State Trait Anxiety Scale. In addition, for the diagnosis of urinary tract infection in participants undergoing CIC, urinalysis will be performed once a month, three times for three months. Patients with 100,000 colonies per milliliter of urine for urinalysis will be considered to have a urinary tract infection. No additional intervention will be made to caregivers in the control groups. Caregivers in the intervention group (Caregivers who will receive CIC training supported by Android phone application based on Roy adaptation model) will be given CIC training, home visit, and telephone conversation. In addition, an android phone application will be installed on the phones of the caregivers in the intervention group, which reminds the CIC times, procedure steps and hospital appointments. The data will be analyzed using SPSS versiyon with descriptive statistics, Independent t test and Anova in repeated measurements p<0.05 will be statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being literate
* Having a smart phone with an android application
* He should not have received information from the nurse about CIC application.

The children included in our research;

* Between the ages of 0-17
* Karadeniz Technical University Farabi Hospital Pediatric Nephrology Department decided to apply and implement CIC
* It should not have a complex congenital anatomical anomaly of the urogenital system

Exclusion Criteria:

* Being 18 years old and above
* Being a communication problems
* Having mental confusion or any psychiatric problem caregiver
* Not volunteering to participate in the research
* Not have androıd smart phone

Ages: 27 Days to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participants are 9 boys and 31 girls. While randomization, grouping was made according to gender. 4 of the boys were in the experimental group and 5 were in the control group.
Enrollment: 40 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2021-05-25 (Estimated)

PRIMARY OUTCOMES:
knowledge / skill level of caregivers. | Change from knowledge / skill level of caregivers at 3 months
  The data collection tool used is not a scale. Created by researchers in line with the literature
The coping / adaptation scala of the caregivers. | Change from the coping / adaptation level of caregivers at 2 months
  Çatal in 2015. The Coping and Adaptation Processing Scale (CAPS) is a 47-item instrument using a Likert scale format with response choices ranging from 4 (always) to 1 (never). Each item of the CAPS is a short statement about how an individual responds to experiencing a crisis or extremely difficult event. Fourteen items are reversed scored. The possible range of scores is from 47 to 188 with a high score indicating a more consistent use of the identified strategies of coping.
Anxiety Level of caregivers | Change from anxiety level of caregivers at 2 months
  State and Trait Anxiety Scale (STAI) will be used to assess the anxiety levels of caregivers. The scale was created in 1964 by Speilberger and Gorsuch. The scale was adapted to Turkish in 1975 by Öner and Le Compte. The scale consists of two parts, each consisting of 20 items. the first part is the state anxiety scale part. Grouped as (1) None, (2) A little, (3) Much, and (4) All. There are ten reversed statements in the state anxiety scale. These are Articles 1, 2,5, 8, 10, 11, 15, 16, 19 and 20. Trait Anxiety Scale is the second part of the scale. Grouped as (1) Almost never, (2) Sometimes, (3) A lot of time, and (4) Almost always. Reversed on the trait anxiety scale there are expressions. These statements are 21, 26, 27, 30, 33, 36 and 39. The scores obtained from each scale range from 20 to 80. The higher the scores obtained from the scale, the higher the anxiety level.
Urinary infection in the child. | Change from Urinary infection in the child at 2 months
  Urine analysis will be performed to evaluate the development of urinary tract infection in children undergoing CIC.The diagnosis of urinary tract infection in children will be made in accordance with the literature with the presence of 100,000 colony bacteria in the urine.
Roy adaptatıon model question form | Change from at 2 months
  Question form created by adhering to NANDA-I nursing diagnoses based on the concepts in the Roy Adaptation Model and the stimuli in the model.The data collection tool used is not a scale. Created by researchers in line with the literature

CONTACTS AND LOCATIONS:
Overall Officials: CANAN SARI, PhD student, Principal Investigator — Karadeniz Technical University
Locations (2):
- Turkey (Türkiye) (2):
  - Karadeniz Techical University Health Faculty of Health Sciences, Trabzon, Health Faculty of Health Sciences
  - Karadeniz Technıcal University, Trabzon, Health Faculty of Health Sciences

IPD SHARING:
Plan to Share IPD: No
I do not want to share my individual participant data with other participants, as I have not completed my work yet.

REFERENCES:
- [Result] Gould CV, Umscheid CA, Agarwal RK, Kuntz G, Pegues DA; Healthcare Infection Control Practices Advisory Committee. Guideline for prevention of catheter-associated urinary tract infections 2009. Infect Control Hosp Epidemiol. 2010 Apr;31(4):319-26. doi: 10.1086/651091. No abstract available. PMID 20156062
- [Result] Lapides J, Diokno AC, Gould FR, Lowe BS. Further observations on self-catheterization. J Urol. 1976 Aug;116(2):169-71. doi: 10.1016/s0022-5347(17)58730-3. PMID 950697
- [Result] Singh R, Rohilla RK, Sangwan K, Siwach R, Magu NK, Sangwan SS. Bladder management methods and urological complications in spinal cord injury patients. Indian J Orthop. 2011 Mar;45(2):141-7. doi: 10.4103/0019-5413.77134. PMID 21430869
- [Result] Neveus T, von Gontard A, Hoebeke P, Hjalmas K, Bauer S, Bower W, Jorgensen TM, Rittig S, Walle JV, Yeung CK, Djurhuus JC. The standardization of terminology of lower urinary tract function in children and adolescents: report from the Standardisation Committee of the International Children's Continence Society. J Urol. 2006 Jul;176(1):314-24. doi: 10.1016/S0022-5347(06)00305-3. PMID 16753432
- [Derived] Sari C, Demirbag BC. The effect of model-based android phone application supported clean intermittent catheterization training on caregivers and children: A randomized controlled study. Eur J Pediatr. 2024 Nov 27;184(1):46. doi: 10.1007/s00431-024-05890-z. PMID 39601932